CLINICAL TRIAL: NCT04463199
Title: Effects of Deep Cervical Flexors Training On Forward Head Posture, Neck Pain and Functional Status in Adolescent Children Using Computer Regularly
Brief Title: Effects of Deep Cervical Flexors Training On Forward Head Posture, Neck Pain and Functional Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRC-2019-08
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Forward Head Posture; Neck Pain
Keywords: Neck pain; Forward head posture; Deep cervical flexors
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental group received craniocervical flexion training for 4 weeks and postural advice
  Interventions: Other: Craniocervical flexion training
- Control Group (No Intervention): Control group received only postural advice

INTERVENTIONS:
Other: Craniocervical flexion training — PBU airbag was clipped together and folded in, fastened, and placed suboccipital. Uninflated pressure sensor was kept below the neck, so that it touched the occiput then inflated to a stable baseline pressure of 20 mmHg to just fill the space below the neck but not to push it into lordosis. Subjects were demonstrated the correct action of the deep cervical flexors that is gentle nodding of head as if saying "yes".
  Arms: Experimental

SUMMARY:
Using computer for long hours is related to higher risk of computer related muscular disorders like forward head posture and neck pain. Deep cervical flexor muscles are important head-on-neck posture stabilizers thus their training may lead to improvement in forward head posture (FHP) and neck pain (NP).

DETAILED DESCRIPTION:
In contemporary societies, computer use by children is a necessity and thus highly prevalent. Using computer for long hours is related to higher risk of computer-related muscular disorders like forward head posture and neck pain. Deep cervical flexor muscles are important head-on-neck posture stabilizers thus their training may lead to improvement in forward head posture (FHP) and neck pain (NP). Aim of study was to determine if 4 weeks of deep cervical flexors training is effective in alleviating neck pain and improving forward head posture in adolescent children using computer regularly. A pretest-posttest experimental group design was used. Subjects were randomly assigned into control group (receiving postural advice only) and experimental group (receiving deep cervical flexor training and postural advice). Dependent variables were measured on day 0 (at baseline) and after 4weeks of training. The photographic analysis was used for measuring forward head posture, visual analog scale (VAS) for neck pain intensity and Neck Disability Index (NDI) for functional disability. Experimental group received craniocervical flexion training for 4 weeks and postural advice. Control group received only postural advice.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain with or without headache, of duration more than 3 months and less than 1 year and 6 months, as identified by body discomfort chart and
* Neck disability index value less than 24 (mild to moderate disability scores on NDI)
* Forward head posture as identified by straight line down from external meatus falling anterior to shoulder and mid thorax.
* Using computer for at least 3 hours a day for at least 4 days a week or more.

Exclusion Criteria:

* Ongoing or previous history of spinal fracture
* Ongoing or previous history of neurological signs
* Ongoing or previous history of inflammatory disease
* Ongoing or previous history of spinal tumor
* Ongoing or previous history of spinal infection
* Ongoing or previous history of spinal cord compression
* Ongoing or previous history of congenital, or acquired postural deformity
* Ongoing or previous history of cervical spinal surgery
* Ongoing or previous history of spinal instability

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Change in craniovertebral angle | 4 weeks
  Change in the craniovertebral angle is assessed from baseline at 4 weeks interval.

SECONDARY OUTCOMES:
Change in Neck Disability Index | 4 weeks
  Change in Functional status is assessed from baseline at 4 weeks interval.
Change in Visual Analog Scale | 4 weeks
  Change in Neck pain intensity assessed from baseline at 4 weeks interval. It is a scale on a piece of paper equal to the length of 10 cm. Each centimeter has 1 point, with 0 means "no pain" and 10 means "worst pain felt ever". Lower the score, better the outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided